CLINICAL TRIAL: NCT04707144
Title: Performance Evaluation of a 3D PSIR Sequence in MRI at 1.5T in the Detection and Characterization of Spinal Cord Injuries in Patients With Multiple Sclerosis
Brief Title: Performance Evaluation of a 3D PSIR Sequence in MRI at 1.5T
Acronym: ESPOIR1-5
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: ALR_2020_40
Record Dates: First submitted 2021-01-11; First posted 2021-01-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: MRI 1.5 tesla — * standard imaging protocol prescribed as part of the usual treatment: sagittal T1 and T2 slices after injection of contrast product (Gadolinium), o 3D STIR sequence.
  * 3D PSIR sequence at the level of the cervical cord for the duration of the additional sequence is 10 minutes, for a total examination time of 45 minutes (instead of 35 minutes)

SUMMARY:
Inclusion visit (D0):

* verification of inclusion and non-inclusion criteria
* information and collection of consent
* standard imaging protocol prescribed as part of the usual treatment: sagittal T1 and T2 slices after injection of contrast product (Gadolinium), o 3D STIR sequence.
* 3D PSIR sequence at the level of the cervical cord for the duration of the additional sequence is 10 minutes, for a total examination time of 45 minutes (instead of 35 minutes).

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old
* To benefit from a medullary exploration planned by MRI 1.5T as part of a first evaluation or a re-evaluation of inflammatory involvement of the nevrax
* Express consent to participate in the study
* Affiliate or beneficiary of a social security scheme

Exclusion Criteria:

* Patient benefiting from a legal protection measure
* Pregnant, parturient or breastfeeding woman
* Absolute or relative contraindication to MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be offered prospectively to patients presenting to the imaging department for a 1.5T MRI for bone marrow exploration, in the context of inflammatory involvement of the nevrax
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2021-05-06 (Actual); Primary Completion 2023-06-06 (Actual); Study Completion 2023-06-28 (Actual)

PRIMARY OUTCOMES:
Estimate the number of spinal cord injuries detected with the set of standard sequences (T1, T2 and STIR) that are not detected with the 3D PSIR sequence | 1 DAY
Estimate the number of active lesions taking the contrast after injection of gadolinium, with the 3D PSIR sequence which is not detected in the set of standard sequences (T1, T2 and STIR) | 1 day
Compare the diagnostic confidence expressed by the radiologist for the detection of spinal cord injuries with the 3D PSIR sequence compared to the set of standard sequences (T1, T2 and STIR) | 1 DAY
Describe the quality of the images in terms of artifacts for each of the sequences used (T1, T2, STIR and PSIR) | 1 DAY
Measure the signal-to-noise ratio of each of the sequences used (T1, T2, STIR and PSIR) | 1 DAY
Measure the inter-observer agreement on the number of lesions detected with the 3D PSIR sequence | 1 DAY
Measure the intra-observer agreement on the number of lesions detected with the 3D PSIR sequence | 1 DAY

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - CHU DE Bordeaux, Bordeaux
  - Chu de Clermont-Ferrand, Clermont-Ferrand
  - Chu de Lille, Lille
  - CHU de LYON, Lyon
  - Hôpital privé des Peupliers, Paris
  - Fondation Ophtalmologique Adolphe de Rothschild (FOR), Paris